CLINICAL TRIAL: NCT06629168
Title: Usage of Telemetric Prechamber Sensor Reservoir in Management of Hydrocephalus
Brief Title: The Usage of Telemetric Prechamber Sensor Reservoir in Management of Normal Pressure Hydrocephalus. Comparisson of Benefit for Patients with Implanted Telemetric Prechamber Sensor Reservoir.
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Miroslav Cihlo, Principal Investigator, University Hospital Hradec Kralove
Other Study IDs: MC00003
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Hydrocephalus; Normal Pressure Hydrocephalus; Normal Pressure Hydrocephalus Patients
Keywords: Normal pressure hydrocephalus; VP drainage; telemetry; pressure monitoring
MeSH Terms: conditions — Hydrocephalus; Hydrocephalus, Normal Pressure | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group "Telemetrics": Patients with diagnosed hydrocephalus undergoing surgery (VP shunt placement) in general anesthesia. During surgery telemetrical prechamber implantad.
  Interventions: Diagnostic Test: lumbar puncture; Diagnostic Test: External lumbar drainage; Procedure: Ventriculo-peritoneal shunt placement; Diagnostic Test: Follow-up control #1; Diagnostic Test: Follow-up control #2; Diagnostic Test: Follow-up control #3; Diagnostic Test: Follow-up control #4; Diagnostic Test: Telemetric prechamber reading; Other: Valve setting change
- Study group "Normal": Patients with diagnosed hydrocephalus undergoing surgery (VP shunt placement) in general anesthesia. During surgery telemetrical prechamber not implantad.
  Interventions: Diagnostic Test: lumbar puncture; Diagnostic Test: External lumbar drainage; Procedure: Ventriculo-peritoneal shunt placement; Diagnostic Test: Follow-up control #1; Diagnostic Test: Follow-up control #2; Diagnostic Test: Follow-up control #3; Diagnostic Test: Follow-up control #4; Other: Valve setting change

INTERVENTIONS:
Diagnostic Test: lumbar puncture — Standardized lumbar puncture in L3/4 or L4/5 in diagnosis of hydrocephalus and 10-meter-walking test prior and 4 hours after lumbar puncture. Mini-mental state examination is done.
Diagnostic Test: External lumbar drainage — External lumbar drainage placement for assessing responsivity of external derivation of cerebrospinal fluid. It is test of responsivity to ventriculo-peritoneal shunt placement
Procedure: Ventriculo-peritoneal shunt placement — Surgical procedure based on implantation a thin catheter into brain lateral ventricle (placed through a burrhole from Kocher point) and connection to prechamber and valve (placed behind the ear under skin) and similar thin catheter pushed under skin of neck, chest and abdomen (where put intraperitoneally). Telemetric prechamber placement according the randomization (www.randomization.com) and the envelope method of choosing of patients.
Diagnostic Test: Follow-up control #1 — Patients after VP shunt placement are assesed in gait, general condition and mini-mental state examination score 3 month after surgery. Brain CT control.
Diagnostic Test: Follow-up control #2 — Patients after VP shunt placement are assesed in gait, general condition and mini-mental state examination score 6 month after surgery. Brain CT control.
Diagnostic Test: Follow-up control #3 — Patients after VP shunt placement are assesed in gait, general condition and mini-mental state examination score 9 months after surgery. Brain CT control.
Diagnostic Test: Follow-up control #4 — Patients after VP shunt placement are assesed in gait, general condition and mini-mental state examination score a month after surgery. Brain CT control, 10-meter-walking test, MMSE, self-assessment.
Diagnostic Test: Telemetric prechamber reading — Non-invasive reading of telemetric prechamber made during each follow-up control.
  Groups: Study group "Telemetrics"
Other: Valve setting change — Changing of valve setting according patient's actual condition. Decission based on clinical state, radiological finding on CT and values readed from telemetric prechamber. Timing - each follow-up control.

SUMMARY:
Normal pressure hydrocephalus (NPH) is a preventable and treatable cause of dementia. However, as a nosological entity, it is significantly underdiagnosed, often being mistakenly classified as presenile or senile dementia without further investigation. Ongoing management is crucial, currently relying mainly on indirect methods-clinical and imaging-based. Telemetry offers a real-time, online method to assess actual cerebrospinal fluid pressures, which are crucial for patient management. Telemetry allows for tailoring treatment to the individual patient. This project is planned as a pilot study before a more extensive research project.

DETAILED DESCRIPTION:
Normal pressure hydrocephalus (NPH) is a preventable and treatable cause of dementia. However, as a nosological entity, it is significantly underdiagnosed, often being mistakenly classified as presenile or senile dementia without further investigation. Diagnosing NPH is not straightforward; it is based on a series of examinations, the results of which determine whether the patient is a responder and therefore a candidate for shunt surgery (implantation of a ventriculoperitoneal shunt). The medical literature identifies additional criteria that predict whether the implantation of the shunt will have a good or poor effect. However, treatment from a neurosurgical perspective does not end there. Ongoing management is crucial, currently relying mainly on indirect methods-clinical and imaging-based. Telemetry offers a real-time, online method to assess actual cerebrospinal fluid pressures, which are crucial for patient management. Telemetry allows for tailoring treatment to the individual patient. This project is planned as a pilot study before a more extensive research project.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed communicating hydrocephalus
* mini-mental state examination test > 10 points
* Absence of any structural lesion on MRI or CT
* Accepted Informed consent

Exclusion Criteria:

* Non-communicating hydrocephalus
* Structural lesion on MRI or CT (tumour, contusion, aneurysm)
* mini-mental state examination test < 10 points
* Life-expectancy shorter than 1 year
* Pre-existing other type of dementia (m. Alzheimer, vascular dementia)
* Surgery lasting more than 120 minutes
* Blood loss more than 500 ml
* Adverse events during general anesthesia: mean arterial pressure < 60 mm Hg more than 5 minutes, arrythmia with need for pharmacological treatment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected based on inclusion criterias, with communicating hydrocephalus
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of patient's state | 3 month
  Comparison of mini-mental state examination, gait (measured by 5-meter-walking) test a self-assessment made by patient between both group (telemetric prechamber impanted versus not implanted)

SECONDARY OUTCOMES:
Comparison in radiological findings | 1 year
  Comparison of size of brain ventricles on brain CT examination at the end of follow-up between both groups
Comparison in number of valve setting | 1 year
  Comparison in number of valve setting between both groups
Comparison of difference in valve settings | 1 year
  Comparison of difference in valve settings - between pressure set in time of implantation and at the end of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Cihlo, M.D., Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia